CLINICAL TRIAL: NCT04642196
Title: COVID-19 in Home Healthcare and Mortality
Brief Title: COVID-19 in Home Healthcare
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Lena Nilsson, Dr, University Hospital, Linkoeping
Other Study IDs: Home healthcare 2020
Record Dates: First submitted 2020-11-22; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of cause of Death in home Healthcare residents in Östergötland County, Sweden, who had a positive COVID-19 diagnosis and died between March and September 2020.

Our aim is to evaluate the pattern of comorbidity and frailty in a group of individuals in home healthcare with positive COVID-19 diagnoses who had a fatal outcome, and a second aim is to assess the contribution of COVID-19 to those fatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult (< 18 years) individuals and
* cared for in home healthcare in Östergötland county and
* positive COVID-19 diagnosis and
* diseased between March and September 2020

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult residents in home health care.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Frailty | Up to one month before death
  Frailty is classified i four groups:
  * None or mild frailty: no restrictions in daily life.
  * Moderate frailty: mobile and independent but unable to handle physically demanding activities or work.
  * Considerable frailty: able to perform activities of daily living but confined at times to bed or chair.
  * Severe frailty: unable to perform activities of daily living and/or confined to bed or chair. Dementia necessitating care.
Comorbidity | Up to one month before death
  Comorbidity is classified in three Groups: none or mild comorbidity (0-1 diagnosis), moderate comorbidity (2 diagnoses), and severe comorbidity (3 or more diagnoses)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of anesthesia, Linköping, Sweden

REFERENCES:
- [Derived] Nilsson L, Andersson C, Sjodahl R. COVID-19 as the sole cause of death is uncommon in frail home healthcare individuals: a population-based study. BMC Geriatr. 2021 Apr 20;21(1):262. doi: 10.1186/s12877-021-02176-z. PMID 33879078